CLINICAL TRIAL: NCT01911260
Title: Effect of Weekly Zinc Chelate Supplementation on Schoolchildren's Growth: a Randomized Double-blind Controlled Trial
Brief Title: Weekly Zinc Chelate Supplementation on Children's Growth
Acronym: APZinc
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Ana Paula Poblacion, Master in Science, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: APoblacionZinc
Record Dates: First submitted 2013-06-27; First posted 2013-07-30 (Estimated); Results first posted 2013-12-24 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-11

CONDITIONS: Short Stature
Keywords: Zinc; Growth; Child; Dietary Supplements; Randomized Controlled Trial
MeSH Terms: conditions — Dwarfism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Growth Deficit+zinc amino acid chelate (Active Comparator): Children with one and a half or more standard deviations below the mean height for age and gender of the reference population (Z-score under -1.6) were included in the Growth Deficit group (GD).
  During twelve weeks, children received weekly 1ml of lemon flavor caramel syrup containing zinc amino acid chelate at 3%, i.e. the equivalent to 30mg of elemental zinc per ml, disposed into an individual amber glass, containing 20ml of syrup. The supplement administration was made individually with 1ml BD Plastipak disposable syringe, directly into the child's mouth, by the principal investigator. The chosen supplementation day was Tuesday. Therefore, the following weekdays were reserved to supplement any absent student.
  Interventions: Dietary Supplement: Zinc amino acid chelate
- Growth Deficit receiving placebo (Placebo Comparator): Children with one and a half or more standard deviations below the mean height for age and gender of the reference population (Z-score under -1.6) were included in the Growth Deficit group (GD).
  During twelve weeks, children received weekly 1ml of lemon flavor caramel syrup, disposed into an individual amber glass, containing 20ml of syrup. The supplement administration was made individually with 1ml BD Plastipak disposable syringe, directly into the child's mouth, by the principal investigator. The chosen supplementation day was Tuesday. Therefore, the following weekdays were reserved to supplement any absent student.
  Interventions: Other: Placebo
- Normal Height receiving placebo (Placebo Comparator): For the Normal Stature group (NS), HAZ was set up as being between -1 and +1 standard deviations from the mean height reference for age and sex.
  During twelve weeks, children received weekly 1ml of lemon flavor caramel syrup, disposed into an individual amber glass, containing 20ml of syrup. The supplement administration was made individually with 1ml BD Plastipak disposable syringe, directly into the child's mouth, by the principal investigator. The chosen supplementation day was Tuesday. Therefore, the following weekdays were reserved to supplement any absent student.
  Interventions: Other: Placebo
- Normal Height+zinc amino acid chelate (Active Comparator): For the Normal Stature group (NS), HAZ was set up as being between -1 and +1 standard deviations from the mean height reference for age and sex.
  During twelve weeks, children received weekly 1ml of lemon flavor caramel syrup containing zinc amino acid chelate at 3%, i.e. the equivalent to 30mg of elemental zinc per ml, disposed into an individual amber glass, containing 20ml of syrup. The supplement administration was made individually with 1ml BD Plastipak disposable syringe, directly into the child's mouth, by the principal investigator. The chosen supplementation day was Tuesday. Therefore, the following weekdays were reserved to supplement any absent student.
  Interventions: Dietary Supplement: Zinc amino acid chelate

INTERVENTIONS:
Dietary Supplement: Zinc amino acid chelate — During twelve weeks, children received weekly 1ml of lemon flavor caramel syrup containing zinc amino acid chelate at 3%, i.e. the equivalent to 30mg of elemental zinc per ml, disposed into an individual amber glass, containing 20ml of syrup. The supplement administration was made individually with 1ml BD Plastipak disposable syringe, directly into the child's mouth, by the principal investigator. The chosen supplementation day was Tuesday. Therefore, the following weekdays were reserved to supplement any absent student.
  Arms: Growth Deficit+zinc amino acid chelate; Normal Height+zinc amino acid chelate
Other: Placebo — During twelve weeks, children received weekly 1ml of lemon flavor caramel syrup, disposed into an individual amber glass, containing 20ml of syrup. The supplement administration was made individually with 1ml BD Plastipak disposable syringe, directly into the child's mouth, by the principal investigator. The chosen supplementation day was Tuesday. Therefore, the following weekdays were reserved to supplement any absent student.
  Arms: Growth Deficit receiving placebo; Normal Height receiving placebo

SUMMARY:
The purpose of this study is to measure the effect of weekly zinc supplementation on schoolchildren with growth deficit or normal stature.

DETAILED DESCRIPTION:
Zinc is an important micronutrient for humans. Trials with zinc have shown positive effects of supplementation on growth, but there is still a lack of results on schoolchildren population. This Randomized Double-Blind Controlled Trial was design to measure the effect of weekly zinc supplementation on schoolchildren with growth deficit and normal stature. Schoolchildren were allocated into two homogeneous groups named Growth Deficit (HAZ < -1,5 Z-score), and Normal Stature (HAZ between -1,0 and ±1,0 Z-score) and were randomly assigned to compose two exposed and two control groups to receive a supplement of 30mg of zinc amino acid chelate or placebo individually once a week, during 12 weeks. Children's heights were measured at the end of supplementation period and again after 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Children with one and a half or more standard deviations below the mean height for age and gender of the reference population (Z-score under -1.6) were included in the Growth Deficit group (GD). For the Normal Stature group(NS), HAZ was set up as being between -1 and +1 standard deviations from the mean height reference for age and sex.

Exclusion Criteria:

* Children of GD group were evaluated by a Pediatrician specialized in growth disorders with the objective of excluding any organic or genetic condition correlated with growth deficit.

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 199 (Actual)
Dates: Start 2000-09; Primary Completion 2000-12 (Actual); Study Completion 2001-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: José Augusto AC Taddei, MD, Dr PH, Study Director — Federal University of São Paulo

REFERENCES:
- [Derived] Imdad A, Rogner J, Sherwani RN, Sidhu J, Regan A, Haykal MR, Tsistinas O, Smith A, Chan XHS, Mayo-Wilson E, Bhutta ZA. Zinc supplementation for preventing mortality, morbidity, and growth failure in children aged 6 months to 12 years. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD009384. doi: 10.1002/14651858.CD009384.pub3. PMID 36994923

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From original database of 2.519 children, enrolled in the first and second grades of four State-run public basic schools, we selected this study sample using height for age indicator (HAZ). Meetings were held at school with parents/guardians to explain the objective and procedures of the study in order to obtain a written consent.
Pre-assignment Details: From original database (n=2.519), we selected children with one and a half or more standard deviations below the mean height for age (HAZ) and gender of the reference population as Growth Deficit group. For the Normal Height group, HAZ was define as between -1 and +1 standard deviations from the mean height reference for age and sex (n=218).
Groups:
- Growth Deficit + Placebo: Children with one and a half or more standard deviations below the mean height for age and gender of the reference population (Z-score under -1.6) were included in the Growth Deficit group (GD).
  During twelve weeks, children received weekly 1ml of lemon flavor caramel syrup, disposed into an individual amber glass, containing 20ml of syrup. The supplement administration was made individually with 1ml BD Plastipak disposable syringe, directly into the child's mouth, by the principal investigator. The chosen supplementation day was Tuesday. Therefore, the following weekdays were reserved to supplement any absent student.
- Normal Height + Placebo: For the Normal Stature group (NS), HAZ was set up as being between -1 and +1 standard deviations from the mean height reference for age and sex.
  During twelve weeks, children received weekly 1ml of lemon flavor caramel syrup, disposed into an individual amber glass, containing 20ml of syrup. The supplement administration was made individually with 1ml BD Plastipak disposable syringe, directly into the child's mouth, by the principal investigator. The chosen supplementation day was Tuesday. Therefore, the following weekdays were reserved to supplement any absent student.
Period: Supplementation Period
Arm/Group | Growth Deficit+Zinc Amino Acid Chelate | Growth Deficit + Placebo | Normal Height+Zinc Amino Acid Chelate | Normal Height + Placebo
Started | 50 | 50 | 49 | 50
Completed | 40 | 38 | 39 | 42
Not Completed | 10 | 12 | 10 | 8
Not completed — transference or evasion of school | 7 | 9 | 7 | 6
Not completed — Adverse Event | 2 | 0 | 1 | 0
Not completed — refused to receive supplement | 1 | 0 | 1 | 0
Not completed — less than 12 weeks supplementation | 0 | 3 | 1 | 2
Period: Follow-up Period
Arm/Group | Growth Deficit+Zinc Amino Acid Chelate | Growth Deficit + Placebo | Normal Height+Zinc Amino Acid Chelate | Normal Height + Placebo
Started | 40 | 38 | 39 | 42
Completed | 27 | 18 | 24 | 30
Not Completed | 13 | 20 | 15 | 12
Not completed — transference or evasion of school | 13 | 20 | 15 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Growth Deficit+Zinc Amino Acid Chelate | Growth Deficit + Placebo | Normal Height+Zinc Amino Acid Chelate | Normal Height + Placebo | Total
Number analyzed (Participants) | 50 | 50 | 49 | 50 | 199
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 50 | 50 | 49 | 50 | 199
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 7.63 (0.66) | 7.64 (0.71) | 7.63 (0.66) | 7.64 (0.71) | 7.63 (0.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 24 | 25 | 99
  Male | 25 | 25 | 25 | 25 | 100
Region of Enrollment [Number; unit: participants]
  Brazil | 50 | 50 | 49 | 50 | 199

OUTCOME MEASURES:

1. Primary Outcome: Change in Height-for-Age Z-score (HAZ) From End of Supplementation to End of Follow-up Period.
Description: Schoolchildren were allocated into two homogeneous groups named Growth Deficit (HAZ < -1,5 Z-score), and Normal Height (HAZ between -1,0 and ±1,0 Z-score), and were randomly assigned to compose two exposed groups to receive a supplement of 30mg of zinc amino acid chelate, and two control groups to receive placebo individually once a week, during 12 weeks. Children's heights were measured at the End of Supplementation period and again after 12 weeks (Follow-up period). In combination with sex and age we transformed stature to Height-for-Age, expressed in Z-score, which was calculated as a number of standard deviations or Z-scores below or above the reference mean or median value, according to the formula below:
  Z-score = (observed value - median value of the reference population) / standard deviation value of reference population.
  We analyzed and discussed the change in HAZ (HAZ at the End of Follow-up period - HAZ at End of Supplementation).
Time Frame: Height-for-Age Z-score was measured at the End of Supplementation period and again at the End of Follow-up period, with a 12 weeks interval.
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | Growth Deficit+Zinc Amino Acid Chelate | Growth Deficit + Placebo | Normal Height+Zinc Amino Acid Chelate | Normal Height + Placebo
Number analyzed (Participants) | 27 | 18 | 24 | 30
Z-Score | 0.04 (0.12) | -0.08 (0.45) | 0.10 (0.15) | 0.02 (0.26)
Statistical Analysis 1: Comparison: Growth Deficit+Zinc Amino Acid Chelate vs Growth Deficit + Placebo; Null Hypothesis: There isn't difference in the HAZ mean difference between children with Growth Deficit who received zinc amino acid or placebo. We attributed α=0.05, β=0.20, and power=0.80; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; In intragroup of supplementation (zinc or placebo) we used the t-test for dependent samples in order to compare growth over time; Mean Difference (Final Values) = 0.12, Standard Deviation 2.0
Statistical Analysis 2: Comparison: Normal Height+Zinc Amino Acid Chelate vs Normal Height + Placebo; Null Hypothesis: There isn't difference in the HAZ mean difference between children with Normal Height who received zinc amino acid or placebo. We attributed α=0.05, β=0.20, and power=0.80; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.08, Standard Deviation 2.0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during 12 weeks.
Description: In the collection data spread sheet, there was a column for side effects (yes/no), and type of side effects (description given by the subject).
Arm/Group | Growth Deficit+Zinc Amino Acid Chelate | Growth Deficit Receiving Placebo | Normal Height+Zinc Amino Acid Chelate | Normal Height Receiving Placebo
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/49 | 0/50
Other Adverse Events (participants affected / at risk) | 2/50 | 0/50 | 1/49 | 0/50
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Growth Deficit+Zinc Amino Acid Chelate (N=50) | Growth Deficit Receiving Placebo (N=50) | Normal Height+Zinc Amino Acid Chelate (N=49) | Normal Height Receiving Placebo (N=50)
Gastrointestinal event (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The sample loss is a factor that hinders the adoption of results as definitive. Even if they remained similar according to biodemographic variables, we cannot guarantee the maintenance of group equality defined in randomization.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No